CLINICAL TRIAL: NCT02342912
Title: Translation of Social Media Obesity Treatment Into Two College Campus Communities
Brief Title: Social Media Obesity Treatment for College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: University of Massachusetts, Boston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK100916 (NIH)
Record Dates: First submitted 2014-12-16; First posted 2015-01-21 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2019-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Social Media Targeted Treatment (Experimental): Participants randomly assigned to this treatment arm will receive weight loss materials via text messages, Facebook postings, on-line videos, and weekly reports. The topics relate to relate to behavioral and lifestyle changes associated with weight-loss (e.g., nutrition, exercise, social support, and self-monitoring). Calorie and physical activity targets also are set. Participants will receive a suggestion to track diet, physical activity, and weight.
  Interventions: Behavioral: Social Media Treatments
- Social Media Tailored Treatment (Experimental): Participants randomly assigned to this treatment arm receive all of the same weight loss materials (as well as weight, calorie, and physical activity targets) as the Targeted group above. Weekly reports will be more personalized to help participants track diet, physical activity, and weight. Additionally, participants will be asked to report on their weight, exercise and calorie goals, and receive feedback.
  Interventions: Behavioral: Social Media Treatments
- Social Media Contact Control (Active Comparator): Participants randomly assigned to this treatment arm receive health information via text messages, Facebook postings, on-line videos, and weekly reports. Topics relate to having a healthy body weight through a healthy mind, body, and energy. Some topics include stress management, importance of sleep, and importance of accepting one's body. Participants will receive a suggestion to track stress, body image, and energy levels.
  Interventions: Behavioral: Social Media Treatments

INTERVENTIONS:
Behavioral: Social Media Treatments — Each of the three intervention groups offers information that has been shown to be important for college students to have a healthy body weight. All three groups provide information on topics that we know are related to having a healthy body weight, like managing stress, keeping track of how you spend your time, and increasing self-awareness of certain health behaviors. Two of the three programs are focused on weight loss for a healthy body. The third group focuses on having a healthy mind, body and having energy during college.

SUMMARY:
This is a randomized trial designed to translate and deliver programs via social media for a healthy body weight to university students. Specifically, in this trial, we will randomly assign 450 overweight/obese (BMI between 25-45kg/m2) university students (ages 18-35) enrolled at two colleges (George Washington University and University of Massachusetts-Boston) to one of two social media weight loss treatments (personalized or generic) or a contact control. The social media treatments consist of Facebook groups to provide social support, connectedness and intervention content, as well as daily text messages. Assessments will be conducted at baseline, 6, 12, and 18 months post baseline, with the primary outcome being weight loss at 18 months. We hypothesize that: a) Tailored Social Media will lose significantly more weight at the above time points compared with Targeted Social Media. b) Both the Tailored Social Media and Targeted Social Media groups will have greater weight loss at the 6, 12, 18 month follow-ups than Contact Control. The secondary aim is to evaluate changes in metabolic risk factors among those participants who have maintained at least 5% weight loss at 18 months. We hypothesize that participants who achieve a 5% weight loss at 6 and 18 months will have significantly lower triglycerides, higher HDL cholesterol, and lower blood pressure than those who do not achieve and maintain that weight target. Finally, we will conduct additional formative work to evaluate the implementation feasibility of this intervention on college campuses, including an assessment of costs as well as the sustainability infrastructure using the PRISM (Practical, Robust Implementation and Sustainability Model) model as a guide. The results of this study have the potential to significantly impact the delivery of obesity treatment services on college campuses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 35 years old
2. BMI between 25 and 45
3. Current student at GWU, UMB, or other approved college/university in the greater DC/Boston area available for assessments at months 6, 12 and 18
4. Fluent in English
5. Active Facebook user, as identified by current Facebook account, logged in at least one time in the past month
6. Regular text message access

Exclusion Criteria:

1. Untreated hypertension, hyperlipidemia, or type 2 diabetes, unless permission is provided by their health care provider. During screening visits, blood pressure will be assessed. Individuals with blood pressure levels >140/90 mmHg, will be informed of these levels and recommend that they contact their HCP. Study participation cannot commence or resume without HCP consent Note: Since weight control is an appropriate initial treatment for these medical issues, individuals can participate in the trial if they receive permission from their HCP, and the HCP indicates that he/she will be managing these risk factors. Participants who do not currently have a HCP will be connected with Student Health Services on each campus.
2. Heart disease, heart problems, or participants who report being prescribed drugs for blood pressure or a major heart condition, unless permission is received from their HCP. [PAR-Q]
3. Health problems which may influence the ability to walk for physical activity (e.g., chest pain during periods of activity, loss of consciousness or losing balance due to dizziness) or other reasons why a person should not do physical activity, unless permission is provided by their HCP. [PAR-Q]
4. Type 1 diabetes or treatment of type 2 diabetes with insulin or oral medications that may cause hypoglycemia (e.g. sulphonylureas). These individuals will be excluded to mitigate concerns about hypoglycemia in a weight loss program.
5. Health problems that may be associated with unintentional weight change or affect the safety of a weight loss program:

   * Report of a heart attack or stroke
   * Active tuberculosis
   * HIV
   * Chronic hepatitis B or C, or other chronic liver disease
   * Inflammatory bowel disease requiring treatment within the 12 months
   * Thyroid disease
   * Renal disease
   * Hospitalization for asthma or other lung disease in the past year
   * Chronic use of steroid medication.
   * Cancer within the past 5 years (except for non-melanoma skin cancers or early stage cervical cancer)
6. Report of a past diagnosis of or treatment for a DSM-V eating disorder (anorexia nervosa, bulimia nervosa, or binge eating disorder) or meet criteria as based on EDDS screening at start of trial
7. Report of a past diagnosis of or current symptoms of alcohol or substance dependence
8. Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months. These individuals may later be re-screened.
9. History of schizophrenia or bipolar disorder ("manic" depression)
10. Hospitalization for depression or other psychiatric disorder within the past 12 months
11. Currently trying to gain weight, or using steroids for muscle mass or weight gain
12. Bariatric (or weight loss) Surgery
13. Participation in another weight loss or physical activity study that would interfere with this study, or taking weight loss medication
14. A member of a participant's self-identified close social network is a participant
15. If graduate student, being in a support or evaluative role of undergraduate students on same campus (e.g., resident advisor/director, teaching assistant, coach). If so, this person may be excluded or asked to wait to join a cohort with students from other universities.
16. Reason to suspect that the participant would not adhere to the study intervention or assessment schedule
17. Medications - not stable on dosage for at least 3 months or HCP Clearance depending on medication type.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 18 months
  Magnitude of weight loss among the three study groups
Weight Loss Difference | 18 months
  Mean differences in weight loss among intervention groups compared to control at 18-months post randomization

SECONDARY OUTCOMES:
Metabolic Risk (Change in metabolic risk factors (including blood pressure, total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides) | 18 months
  Change in metabolic risk factors (including blood pressure, total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides) across the three groups and the associated thresholds of weight loss and corresponding metabolic risk.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Napolitano, PhD, Principal Investigator — George Washington University; Jessica A Whiteley, PhD, Study Director — University of Massachusetts, Boston
Locations (2):
- United States (2):
  - The George Washington University, Washington D.C., District of Columbia
  - University of Massachusetts Boston, Boston, Massachusetts

REFERENCES:
- [Derived] Whiteley JA, Tjaden AH, Bailey CP, Faro J, DiPietro L, Hayman LL, Napolitano MA. Engagement with Digital Weight Loss Intervention Components and Weight Outcomes. J Technol Behav Sci. 2024 Dec;9(4):714-723. doi: 10.1007/s41347-024-00388-9. Epub 2024 Feb 3. PMID 41122737
- [Derived] Napolitano MA, Tjaden AH, Bailey CP, DiPietro L, Rimal R. What moves young people? Applying the risk perception attitude framework to physical activity behavior and cardiometabolic risk. Transl Behav Med. 2022 Jul 7;12(6):742-751. doi: 10.1093/tbm/ibac012. PMID 35429404
- [Derived] Napolitano MA, Whiteley JA, Mavredes MN, Faro J, DiPietro L, Hayman LL, Neighbors CJ, Simmens S. Using social media to deliver weight loss programming to young adults: Design and rationale for the Healthy Body Healthy U (HBHU) trial. Contemp Clin Trials. 2017 Sep;60:1-13. doi: 10.1016/j.cct.2017.06.007. Epub 2017 Jun 10. PMID 28611007